CLINICAL TRIAL: NCT01251861
Title: Androgen Receptor Modulation Phase II, Randomized Study of MK-2206 - Bicalutamide Combination in Patients With Rising PSA at High-Risk of Progression After Primary Therapy
Brief Title: Bicalutamide With or Without Akt Inhibitor MK2206 in Treating Patients With Previously Treated Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02648; NCI-2011-02648 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E2809; CDR0000689613; 11-00834; E2809; E2809 (Other: ECOG-ACRIN Cancer Research Group); E2809 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Prostate Carcinoma; Stage I Prostate Cancer AJCC v7; Stage IIA Prostate Cancer AJCC v7; Stage IIB Prostate Cancer AJCC v7; Stage III Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — MK 2206; bicalutamide; Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (observation and bicalutamide) (Active Comparator): Patients undergo observation on weeks 1-12. Patients then receive bicalutamide PO QD on weeks 13-44. Patients with a PSA decline of >= 50% may continue on bicalutamide until week 72 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bicalutamide; Other: Clinical Observation; Other: Laboratory Biomarker Analysis
- Arm B (Akt inhibitor MK2206 and bicalutamide) (Experimental): Patients receive Akt inhibitor MK2206 PO once per week on weeks 1-44 and bicalutamide PO QD on weeks 13-44. Patients with a PSA decline of >= 50% may continue on Akt inhibitor MK2206 and bicalutamide until week 72 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Bicalutamide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK 2206; MK-2206; MK-2206 FREE BASE; MK2206
  Arms: Arm B (Akt inhibitor MK2206 and bicalutamide)
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cassotide; Cosudex; ICI 176,334; ICI 176334; Utamide
Other: Clinical Observation — Undergo clinical observation
  Other Names: observation
  Arms: Arm A (observation and bicalutamide)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving bicalutamide with or without Akt inhibitor MK2206 works in treating patients with previously treated prostate cancer. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as bicalutamide, may lessen the amount of androgens made by the body. Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether bicalutamide is more effective with or without Akt inhibitor MK2206 in treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the two regimens on the proportion of patients with undetectable prostate-specific antigen (PSA) level (< 0.2 ng/mL) at 44 weeks.

SECONDARY OBJECTIVES:

I. To assess the proportion of patients with PSA decline >= 85% at 44 weeks on the combination therapy arm compared to that of bicalutamide monotherapy arm.

II. To assess the distribution of best PSA response in each study arm. III. To assess the time to PSA progression in each arm of the study. IV. To assess the time to PSA nadir in each arm of the study. V. To assess the duration of PSA response in each arm of the study. VI. To characterize the PSA slope pre-study, during treatment, and off treatment.

VII. To evaluate the safety and tolerability of MK-2206 (Akt inhibitor MK2206) in this patient population.

VIII. To determine whether Gleason score has any effect on PSA response to treatment.

IX. To determine whether prior hormonal therapy has any effect on PSA response to treatment.

TERTIARY OBJECTIVES:

I. Samples of the primary tumor specimen will be retrieved for banking and future analysis of the molecular profile of the primary prostate cancer (PC) tissues with emphasis on the androgen receptor (AR) and protein kinase B (Akt) upstream and downstream signaling pathways.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients undergo observation on weeks 1-12. Patients then receive bicalutamide* orally (PO) once daily (QD) on weeks 13-44. Patients with a PSA decline of >= 50% may continue on bicalutamide until week 72 in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive Akt inhibitor MK2206** PO once per week on weeks 1-44 and bicalutamide* PO QD on weeks 13-44. Patients with a PSA decline of >= 50% may continue on MK2206 and bicalutamide until week 72 in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients may begin bicalutamide on weeks 4-11 if the disease worsens.

NOTE: **Patients on Akt inhibitor MK2206 with a PSA < 0.2 ng/mL by week 12 do not receive bicalutamide until PSA rises to >= 0.2 ng/mL.

After completion of study therapy, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then every year for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically confirmed diagnosis of prostate cancer
* Patient must have had previous treatment with definitive surgery or radiation therapy or cryoablation
* Patient may have prior salvage therapy (surgery, radiation or other local ablative procedures) within 4 weeks prior to randomization if the intent was for cure; prophylactic radiotherapy to prevent gynecomastia within 4 weeks prior to randomization is allowed
* Patient must have no evidence of metastatic disease on physical exam, computed tomography (CT) abdomen/pelvis (or magnetic resonance imaging [MRI]), chest x-ray (or CT chest) and bone scan within 8 weeks prior to randomization
* Patient may have had prior neoadjuvant and/or adjuvant therapy (chemotherapy, vaccines or experimental agents) within 4 weeks prior to randomization, if the PSA rise and PSA doubling time (PSADT) were documented after the testosterone level was > 150 ng/dL
* Patient may not have had therapy modulating testosterone levels (such as luteinizing-hormone, releasing-hormone agonists/antagonists and antiandrogens) within 1 year prior to randomization, unless it was in the neoadjuvant and/or adjuvant setting; agents such as 5 alpha reductase inhibitors, ketoconazole, abiraterone, systemic steroids, or herbal supplements known to decrease PSA levels including any dose of megestrol acetate, finasteride (e.g., Saw Palmetto and PC-SPES, African pygeum extract, lycopene, alanine, glutamic acid and glycine, beta-sitosterol, lycopene, nettle root extract, quercitin, Belizian Man Vine extract, mulra puama extract and epimedium extract campesterol, beta-sitosterol, stigmasterol, sitostanol and brassicasterol) are not permitted at any time during the period that the PSA values are being collected
* Patient must have hormone-sensitive prostate cancer as evident by a serum total testosterone level > 150 ng/dL within 12 weeks prior to randomization
* Patient must have evidence of biochemical failure after primary therapy and subsequent progression

  * Biochemical failure is declared when the PSA reaches a threshold value after primary treatment and it differs for radical prostatectomy or radiation therapy
  * For radical prostatectomy the threshold for this study is PSA >= 0.4 ng/mL
  * For radiation therapy the threshold is a PSA rise of 2 ng/mL above the nadir PSA achieved post radiation with or without hormone therapy (2006 Radiation Therapy Oncology Group [RTOG]-American Society for Radiation Oncology [ASTRO] Consensus definition)
  * PSA progression requires a PSA rise above the threshold (PSA1) measured at any time point since the threshold was reached
  * The PSADT must be < 12 months; requires two consecutive PSA rises (PSA2 and PSA3) above the PSA1; PSA2 and PSA3 must be obtained within 6 months of study entry; all baseline PSAs should be obtained, preferably, at the same reference lab
* PSADT calculation needs 3 PSA values:

  * PSA1 is any PSA value that is equal or greater than the threshold PSA (0.4 ng/mL for radical prostatectomy or 2 ng/mL above the nadir for primary radiation therapy) indicating biochemical relapse
  * PSA2 must be higher than PSA1, obtained at least 2 weeks after PSA1 and within 6 months or less from randomization
  * PSA3 must be higher than PSA2 and obtained at least 2 weeks after PSA2
  * Baseline PSA must have reached a minimum of 2 ng/mL but be no greater than 50 ng/mL and equal or higher than PSA3; PSA3 may be used as baseline PSA if obtained within 1 week of randomization
* Patient's PSA doubling time (PSADT) must be less than 12 months
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Granulocytes >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine within normal institutional limits or creatinine clearance >= 50 ml/min for patients with creatinine levels above institutional normal
* Serum total bilirubin =< 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase (ALP) =< 2.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x institutional upper limit of normal
* Human immunodeficiency virus (HIV)-positive patients are excluded from this study
* Patient cannot receive concurrent therapeutic administration of anticoagulant therapy; low dosage aspirin =< 325 mg per day is allowed
* Patients with impaired cardiac function including any one of the following will be excluded from entry on study:

  * Baseline corrected QT interval (QTc) > 450 msec (male) (patients with QTc 450-480 msec will be allowed to participate in this trial if they do not have any of the other cardiac conditions mentioned in this section)
  * Patients with congenital long QT syndrome
  * History of sustained ventricular tachycardia
  * Any history of ventricular fibrillation or torsades de pointes
  * Concomitant use of drugs with a risk of causing torsades de pointes
  * Bradycardia defined as heart rate < 50 beats per minute; patients with a pacemaker and heart rate >= 50 beats per minute are eligible
  * Myocardial infarction or unstable angina within 6 months of study entry
  * Congestive heart failure (New York Heart Association class III or IV)
  * Right bundle branch block and left anterior hemi-block (bifascicular block)
* Patient must not have gastrointestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Patient may not be receiving any other investigational agents or receiving concurrent anticancer therapy (chemotherapy, immunotherapy, radiation therapy, surgery for cancer, or experimental medications) at time of randomization
* Patient may not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 or bicalutamide
* Patient must not have any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with diabetes or at risk for hyperglycemia MUST not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled before the patient enters the trial
* Patients receiving any medications or substances that are inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) are ineligible
* Patient must NOT have previous or concurrent malignancy; exceptions are made for patients who meet any of the following conditions:

  * Basal cell or squamous cell carcinoma of the skin OR
  * Prior malignancy has been adequately treated and patient has been continuously disease free for >= 2 years
* Patient must agree to use barrier contraception during and for 3 months after discontinuation of study treatment; if patient impregnates a woman while on treatment or within 3 months of discontinuing treatment, he should inform his treating physician immediately
* Patients must discontinue use of enzyme-inducing anti-epileptic drugs (EIAEDs) >= 14 days prior to study enrollment; the investigator may prescribe non-EIAEDs; patients who must begin EIAED therapy while on study will be allowed to remain
* Patients must not be taking cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or phenobarbital), St John's Wort, ketoconazole, dexamethasone, the dysrhythmic drugs (terfenadine, quinidine, procainamide, sotalol, probucol, bepridil, indapamide or flecainide), haloperidol, risperidone, rifampin, grapefruit, or grapefruit juice within two weeks of randomization and during the course of therapy
* Patients may have received targeted agents (angiogenesis inhibitors, epidermal growth factor receptor [EGFR] inhibitors, mammalian target of rapamycin [mTOR] inhibitors, phosphatidylinositol 3 kinase [PI3K] inhibitors, etc.), however patients must have discontinued treatment with the targeted agent(s) at least 4 weeks prior to enrollment; if the patient stopped targeted agent(s) due to unresolved or persistent grade 3 or 4 toxicity, patient cannot be enrolled onto the study regardless of the length of time since discontinuation of treatment with targeted agent(s)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-12-23 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2026-03-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anna C Ferrari, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (198):
- United States (192):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Horizon Oncology Research LLC, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Ireland (6):
  - Tallaght University Hospital, Dublin, Co Dublin
  - Saint Vincent's University Hospital, Dublin, Co Dublin
  - Mater Misericordiae University Hospital, Dublin, Co Dublin
  - Mater Private Hospital, Dublin, Co Dublin
  - University College Hospital Galway, Galway, Co Galway
  - Cork University Hospital, Cork

REFERENCES:
- [Derived] Ferrari AC, Chen YH, Rodriguez R, Hudes GR, Antonarakis ES, Hahn NM, Ma H, Plimack ER, Mayer T, Carthon BC, Liu G, Carducci MA, DiPaola R. Phase II Randomized Study of MK-2206 and Bicalutamide in Prostate Cancer Patients With Rising PSA After Primary Therapy (ECOG-ACRIN E2809). Prostate. 2026 Jan 29. doi: 10.1002/pros.70125. Online ahead of print. PMID 41609418

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on December 23, 2010 and closed to accrual on September 20, 2013 with a final accrual of 108 patients from 24 participating sites.
Period: Overall Study
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Started | 54 | 54
Pts Who Received Protocol Therapy | 50 | 53
Pts w/ Follow-up PSA Lower Than Baseline | 49 | 47
Pts With PSA Response | 44 | 36
Completed | 36 | 26
Not Completed | 18 | 28
Not completed — Disease progression | 6 | 6
Not completed — Adverse Event | 2 | 17
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Alternative therapy | 1 | 0
Not completed — Other complicating disease | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Continued treatment beyond 18 cycles | 1 | 0
Not completed — Other | 1 | 0
Not completed — Never started therapy | 4 | 1
Not completed — Potential interaction of drugs | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide) | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Continuous [Median (Full Range); unit: years] | 66 [47 to 81] | 67 [48 to 85] | 66 [47 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 54 | 54 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 50 | 48 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients With Undetectable PSA Level (< 0.2 ng/mL) at 44 Weeks
Description: The proportion of patients with undetectable PSA level (< 0.2 ng/mL) at 44 weeks, defined as number of patients with undetectable PSA level at 44 weeks divided by number of patients randomized.
Time Frame: 44 weeks
Population: All randomized patients are included in this analysis.
Measure: Number (80% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 54 | 54
proportion of participants | 0.093 [0.046 to 0.165] | 0.148 [0.088 to 0.23]
Statistical Analysis 1: Comparison: Arm A (Observation and Bicalutamide) vs Arm B (Akt Inhibitor MK2206 and Bicalutamide); Test type: Superiority; p = 0.28, Fisher Exact — one-sided

2. Secondary Outcome: Proportion of Patients With PSA Decline > 85% at 44 Weeks
Description: Proportion of patients with PSA decline > 85% at 44 weeks from baseline, defined as number of patients with PSA decline > 85% at 44 weeks from baseline divided by number of patients randomized.
Time Frame: 44 weeks
Population: All randomized patients are included in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 54 | 54
proportion of participants | 0.296 [0.18 to 0.436] | 0.426 [0.292 to 0.568]

3. Secondary Outcome: Proportion of Patients With PSA Response
Description: PSA complete response (CR) is defined as a PSA <0.2 ng/mL confirmed on two consecutive additional determinations taken at least 4 weeks apart. PSA partial response (PR) is defined as a reduction in PSA ≥ 50% from baseline without evidence of progression (confirmed on two consecutive additional determinations taken at least 4 weeks apart). Either CR or PR is considered as a PSA response.
Time Frame: Assessed every 3 months for 2 years, every 6 months for 3 years, and then annually up to 10 years
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 54 | 54
proportion of participants | 0.815 [0.686 to 0.908] | 0.667 [0.525 to 0.789]

4. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression was defined as the time from randomization to PSA progression or date of last disease assessment showing progression-free. Development of clinical progression is also considered as an event.
  * For patients (pts) who achieved a ≥ 50% decline in PSA (confirmed on two consecutive determinations taken at least 4 weeks apart), progression is defined as an increase in PSA by 50% above baseline or nadir, whichever is lowest, confirmed by a 2nd PSA rise at least two weeks later. The PSA rise must be >= 5 ng/mL.
  * For pts with an undetectable PSA nadir (< 0.2 ng/mL confirmed on two consecutive determinations taken at least 4 weeks apart), progression is defined as PSA ≥ 0.2 ng/mL confirmed by a 2nd PSA rise at least 2 weeks later.
  * For pts whose PSA has not decreased by 50%, progression is defined as an increase in PSA of ≥ 50% of baseline or nadir PSA, whichever is lowest, confirmed by a repeat PSA at least 2 weeks later. The PSA must have risen by >= 5 ng/mL
Time Frame: Assessed every 3 months for 2 years, every 6 months for 3 years, and then annually up to 10 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 54 | 54
months | 25.8 [21.0 to 37.7] | 24.3 [19.1 to 30.1]

5. Secondary Outcome: Time to PSA Nadir
Description: Time to PSA nadir was defined as the time from randomization to the date that PSA nadir, the lowest PSA value achieved after randomization, was documented. This analysis was performed among patients whose PSA level decreased after randomization compared to baseline.
Time Frame: Assessed every 3 months for 2 years, every 6 months for 3 years, and then annually up to 10 years
Population: Only patients who received protocol therapy and had follow-up PSA level lower than baseline PSA were included.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 49 | 47
months | 7.7 [1.1 to 22.0] | 6.7 [0.3 to 19.3]

6. Secondary Outcome: Duration of PSA Response
Description: Duration of PSA response was defined as the time from the date PSA criteria were met for complete response (CR) or partial response (PR), whichever status was recorded first, to the date of PSA progression. Patients without documented PSA progression were censored at the date of last disease assessment. Duration of PSA response is analyzed among responders (PSA CR or PR).
Time Frame: Assessed every 3 months for 2 years, every 6 months for 3 years, and then annually up to 10 years
Population: Patients with PSA response (CR or PR)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 44 | 36
months | 20.6 [17.0 to 34.7] | 25.3 [17.6 to 37.5]

7. Secondary Outcome: PSA Slope Prior to Randomization
Description: PSA slopes were assessed by multiple PSA values prior to randomization. Linear regression was used to calculate PSA slope using natural log-transformed PSA values on the time of PSA measurements for each patient.
Time Frame: Baseline (pre-randomization)
Population: All randomized patients
Measure: Mean (Standard Deviation); unit: ln(PSA)/month
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 54 | 54
ln(PSA)/month | 0.20 (0.16) | 0.20 (0.13)

8. Secondary Outcome: PSA Slope After Randomization and Before Starting Bicalutamide
Description: PSA slopes were assessed by multiple PSA values from randomization to starting bicalutamide treatment. Linear regression was used to calculate PSA slope using natural log-transformed PSA values on the time of PSA measurements for each patient.
Time Frame: After randomization and prior to starting bicalutamide
Population: Patients with follow-up PSA measurement before starting bicalutamide.
Measure: Mean (Standard Deviation); unit: ln(PSA)/month
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 49 | 53
ln(PSA)/month | 0.10 (0.14) | 0.06 (0.23)

9. Secondary Outcome: PSA Slope After Starting Bicalutamide Treatment
Description: PSA slopes were assessed by multiple PSA values after starting bicalutamide treatment. Linear regression was used to calculate PSA slope using natural log-transformed PSA values on the time of PSA measurements for each patient.
Time Frame: Assessed every 3 months for 2 years, every 6 months for 3 years, and then annually up to 10 years
Population: Patients with follow-up PSA measurement after starting bicalutamide.
Measure: Mean (Standard Deviation); unit: ln(PSA)/month
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 48 | 42
ln(PSA)/month | -0.57 (0.96) | -0.60 (0.57)

10. Secondary Outcome: The Association Between Gleason Score and PSA Response
Description: The association between PSA response (responder vs non-responder) and Gleason score (<7, 7 vs. >7) was evaluated by logistic regression with adjustment for treatment assignment.
  Based on the biopsy sample, a Gleason grade is assigned to the most predominant pattern in the biopsy and a second Gleason grade is assigned to the second most predominant pattern. The two grades will then be added together to determine the Gleason score. Gleason scores range from 2-10. The higher the Gleason score, the more aggressive the cancer is likely to be.
Time Frame: Assessed every 3 months for 2 years, every 6 months for 3 years, and then annually up to 10 years
Population: All randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 54 | 54
Participants
  Gleason score <7: number analyzed (Participants) | 10 | 10
  Gleason score <7: Responder | 9 | 7
  Gleason score <7: Non-responder | 1 | 3
  Gleason score =7: number analyzed (Participants) | 25 | 23
  Gleason score =7: Responder | 20 | 17
  Gleason score =7: Non-responder | 5 | 6
  Gleason score >7: number analyzed (Participants) | 19 | 21
  Gleason score >7: Responder | 15 | 12
  Gleason score >7: Non-responder | 4 | 9
Statistical Analysis 1: Comparison: Arm A (Observation and Bicalutamide) vs Arm B (Akt Inhibitor MK2206 and Bicalutamide); The association between PSA response (responder vs non-responder) and Gleason score (<7, 7 vs. >7) was evaluated by logistic regression with adjustment for treatment assignment; Test type: Other — The association between PSA response (responder vs non-responder) and Gleason score (<7, 7 vs. >7) was evaluated by logistic regression with adjustment for treatment assignment; p = 0.50, Regression, Logistic — p-value based on logistic regression with adjustment for treatment assignment

11. Secondary Outcome: The Association Between Prior Hormonal Therapy and PSA Response
Description: The association between PSA response (responder vs non-responder) and prior hormonal therapy (yes vs. no) was evaluated by logistic regression with adjustment for treatment assignment.
Time Frame: Assessed every 3 months for 2 years, every 6 months for 3 years, and then annually up to 10 years
Population: All randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Observation and Bicalutamide) | Arm B (Akt Inhibitor MK2206 and Bicalutamide)
Number analyzed (Participants) | 54 | 54
Participants
  No prior hormonal therapy: number analyzed (Participants) | 31 | 29
  No prior hormonal therapy: Responder | 28 | 19
  No prior hormonal therapy: Non-responder | 3 | 10
  Received prior hormonal therapy: number analyzed (Participants) | 23 | 25
  Received prior hormonal therapy: Responder | 16 | 17
  Received prior hormonal therapy: Non-responder | 7 | 8
Statistical Analysis 1: Comparison: Arm A (Observation and Bicalutamide) vs Arm B (Akt Inhibitor MK2206 and Bicalutamide); The association between PSA response (responder vs non-responder) and prior hormonal therapy (yes vs. no) was evaluated by logistic regression with adjustment for treatment assignment; Test type: Other — The association between PSA response (responder vs non-responder) and prior hormonal therapy (yes vs. no) was evaluated by logistic regression with adjustment for treatment assignment; p = 0.28, Regression, Logistic — p-value based on logistic regression with adjustment for treatment assignment

12. Other Pre Specified Outcome: Samples of the Primary Tumor Specimen Will be Retrieved for Banking and Future Analysis of the Molecular Profile of the Primary PC Tissues With Emphasis on the AR and Akt Upstream and Downstream Signaling Pathways.
Description: Biospecimen banking for future analysis; no data to be reported
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment (up to about 76 weeks)
Description: All-cause mortality was monitored in all randomized patients and all other adverse events were assessed in participants who received treatment.
Groups:
- Arm A (Observation + Bicalutamide): Patients undergo observation on weeks 1-12. Patients then receive bicalutamide PO QD on weeks 13-44. Patients with a PSA decline of >= 50% may continue on bicalutamide until week 72 in the absence of disease progression or unacceptable toxicity.
- Arm B (MK-2206 + Bicalutamide): Patients receive Akt inhibitor MK2206 PO once per week on weeks 1-44 and bicalutamide PO QD on weeks 13-44. Patients with a PSA decline of >= 50% may continue on Akt inhibitor MK2206 and bicalutamide until week 72 in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (Observation + Bicalutamide) | Arm B (MK-2206 + Bicalutamide)
All-Cause Mortality (participants affected / at risk) | 9/54 | 9/54
Serious Adverse Events (participants affected / at risk) | 1/50 | 33/53
Other Adverse Events (participants affected / at risk) | 39/50 | 52/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Observation + Bicalutamide) (N=50) | Arm B (MK-2206 + Bicalutamide) (N=53)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Blood and lymphatic disorders - Other (Blood and lymphatic system disorders) | 0 | 1
Fatigue (General disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 20
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 5
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 6
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Observation + Bicalutamide) (N=50) | Arm B (MK-2206 + Bicalutamide) (N=53)
Anemia (Blood and lymphatic system disorders) | 3 | 11
Chills (General disorders) | 1 | 3
Edema limbs (General disorders) | 1 | 4
Fatigue (General disorders) | 16 | 33
Fever (General disorders) | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 17
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 24
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 29
Skin and subcutaneous tissue - Other (Skin and subcutaneous tissue disorders) | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 1 | 8
Diarrhea (Gastrointestinal disorders) | 1 | 26
Dry mouth (Gastrointestinal disorders) | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 6
Flatulence (Gastrointestinal disorders) | 0 | 5
Mucositis oral (Gastrointestinal disorders) | 0 | 10
Nausea (Gastrointestinal disorders) | 3 | 10
Alanine aminotransferase increased (Investigations) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 6
Creatinine increased (Investigations) | 2 | 10
Lymphocyte count decreased (Investigations) | 5 | 12
Neutrophil count decreased (Investigations) | 0 | 3
Platelet count decreased (Investigations) | 2 | 8
Weight loss (Investigations) | 0 | 4
White blood cell decreased (Investigations) | 4 | 9
Anorexia (Metabolism and nutrition disorders) | 0 | 10
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 23
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Dizziness (Nervous system disorders) | 1 | 4
Dysgeusia (Nervous system disorders) | 0 | 6
Headache (Nervous system disorders) | 3 | 6
Blurred vision (Eye disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Breast pain (Reproductive system and breast disorders) | 26 | 14
Gynecomastia (Reproductive system and breast disorders) | 21 | 11
Reproductive system and breast - Other (Reproductive system and breast disorders) | 2 | 3
Hot flashes (Vascular disorders) | 11 | 8
Hypertension (Vascular disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/61/NCT01251861/Prot_SAP_000.pdf